CLINICAL TRIAL: NCT00127868
Title: A Randomized, Double-Blinded, Placebo-Controlled Study Observing the Efficacy of Selenium Sulfide 1% Shampoo, Ketoconazole 2% Shampoo, and Ciclopirox 1% Shampoo as Adjunctive Treatments for Tinea Capitis in Children
Brief Title: Selenium Sulfide, Ketoconazole and Ciclopirox Shampoo as Additional Treatments for Tinea Capitis (Scalp Ringworm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen, Catherine, M.D. (Other)
Collaborators: Williams, Judith V., M.D. (Individual); Hubbard, Thomas W., M.D. (Individual); Eastern Virginia Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-Chen
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2006-05

CONDITIONS: Tinea Capitis
Keywords: Tinea Capitis; Children; Pediatric; Treatment; Therapy; Adjunctive; Selenium Sulfide; Ciclopirox; Shampoo
MeSH Terms: conditions — Tinea Capitis | interventions — Griseofulvin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 1 (Active Comparator): oral griseofulvin and selenium sulfide shampoo 1%
  Interventions: Drug: oral griseofulvin, selenium sulfide shampoo 1%, ciclopirox shampoo , ketoconazole shampoo 2%, baby shampoo
- 2 (Active Comparator): oral griseofulvin and ciclopirox shampoo
  Interventions: Drug: oral griseofulvin, selenium sulfide shampoo 1%, ciclopirox shampoo , ketoconazole shampoo 2%, baby shampoo
- 3 (Active Comparator): oral griseofulvin and ketoconazole shampoo 2%
  Interventions: Drug: oral griseofulvin, selenium sulfide shampoo 1%, ciclopirox shampoo , ketoconazole shampoo 2%, baby shampoo
- 4 (Placebo Comparator): oral griseofulvin and baby shampoo
  Interventions: Drug: oral griseofulvin, selenium sulfide shampoo 1%, ciclopirox shampoo , ketoconazole shampoo 2%, baby shampoo

INTERVENTIONS:
Drug: oral griseofulvin, selenium sulfide shampoo 1%, ciclopirox shampoo , ketoconazole shampoo 2%, baby shampoo

SUMMARY:
Antifungal shampoos have been used as supplements to oral griseofulvin to help eradicate tinea capitis (also known as ringworm of the scalp) more quickly. While selenium sulfide shampoo has been the gold standard, its strong odor and its drying effect on the scalp discourage many patients from using it. Meanwhile, no other antifungal shampoo has been rigorously evaluated for efficacy. Therefore, while physicians are prescribing griseofulvin accompanied by any of a number of antifungal shampoos for tinea capitis, it is not known which antifungal shampoos (excluding selenium sulfide) actually significantly reduce time to cure, nor which do so the fastest.

Scalp ringworm can also re-occur in the same child. To date, no studies have been done to find out whether or not the use of antifungal shampoos can prevent the recurrence of scalp ringworm.

In this study, children ages 1-12 years old, who have clinically diagnosed tinea capitis, will all be prescribed oral griseofulvin for 8 weeks. In addition, they will be randomly assigned to use either selenium sulfide shampoo, ketoconazole shampoo, ciclopirox shampoo, or baby shampoo twice a week for 8 weeks. After 8 weeks, griseofulvin will be stopped. All patients will continue using the same assigned shampoo twice weekly for 24 weeks, while continuing to return to clinic every 4 weeks for scalp evaluation.

DETAILED DESCRIPTION:
Antifungal shampoos have been used as supplements to oral griseofulvin to help eradicate tinea capitis (also known as ringworm of the scalp) more quickly. While selenium sulfide shampoo has been the gold standard, its strong odor and its drying effect on the scalp discourage many patients from using it. Meanwhile, no other antifungal shampoo has been rigorously evaluated for efficacy. Therefore, while physicians are prescribing griseofulvin accompanied by any of a number of antifungal shampoos for tinea capitis, it is not known which antifungal shampoos (excluding selenium sulfide) actually significantly reduce time to cure, nor which do so the fastest.

Scalp ringworm can also re-occur in the same child. To date, no studies have been done to find out whether or not the use of antifungal shampoos can prevent the recurrence of scalp ringworm.

In this study, children ages 1-12 years old, who have clinically diagnosed tinea capitis, will all be prescribed oral griseofulvin for 8 weeks. In addition, they will be randomly assigned to use either selenium sulfide shampoo, ketoconazole shampoo, ciclopirox shampoo, or baby shampoo twice a week for 8 weeks. After 8 weeks, griseofulvin will be stopped. All patients will continue using the same assigned shampoo twice weekly for 24 weeks, while continuing to return to clinic every 4 weeks for scalp evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed tinea capitis.
* Males or females, ages 1 through 12 years old.
* Females of childbearing potential must have a negative pregnancy test.
* Written Informed Consent must be obtained prior to performing any study- related procedure and according to local regulations.
* Patients must be available for the entire study duration.

Exclusion Criteria:

* Patients who are pregnant or breast-feeding.
* Patients who have kerions requiring immediate treatment or treatment with systemic corticosteroids and/or systemic antibiotics.
* Patients who have a skin disease involving the scalp, or any other condition or prior/present treatment which in the opinion of the investigator would interfere with evaluation of the treatment's effect. Examples include head lice, scalp psoriasis, atopic dermatitis of the scalp, or seborrheic dermatitis.
* Patients with known liver disease.
* Patients with non-acidic gastroduodenitis, malabsorption syndrome, chronic diarrhea, or any other serious gastrointestinal (GI) disease.
* Patients who have received systemic antifungal treatment within 2 months prior to baseline.
* Patients who have received the following topical treatments for their scalp within 1 week prior to baseline: antifungal agents, corticosteroids, zinc pyrithione, selenium sulfide, or tar-containing products.
* Patients who have received immunosuppressant therapy, cytostatic therapy, or underwent radiation therapy within 1 month prior to baseline.
* Patients who have been treated with any investigational agent within 8 weeks prior to baseline or who intend to use other investigational treatments during this study.
* Patients with hypersensitivity to griseofulvin, selenium sulfide, or ciclopirox.
* Patients who are known to miss appointments (per medical records), unlikely to follow medical instructions, or not willing to attend regular visits.
* The following exclusion criteria are based upon the package insert for griseofulvin microsize suspension:

  * Males planning to father children during their participation in the study or in the 6 months following their completion of the study.
  * Patients taking substances known to interact with griseofulvin.
  * Patients with systemic lupus erythematosus.
  * Patients with porphyria.
  * Patients with photosensitivity.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
efficacy | 9-10 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chen, M.D., Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States